CLINICAL TRIAL: NCT01565967
Title: Registry AutoLog Lipid Removal and Blood Component Characterization
Status: Completed | Type: Observational
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Organization: Medtronic Cardiovascular (Industry)
Other Study IDs: AutoLog
Record Dates: First submitted 2011-06-08; First posted 2012-03-29 (Estimated); Last update posted 2015-10-29 (Estimated); Status verified 2015-10

CONDITIONS: Trauma
Keywords: AutoLog; Post market release; Non-interventional
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood and washed blood will be collected from each patient
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Autotransfusion: All patients undergoing surgery which requires routine use of an autotransfusion system

SUMMARY:
The purpose of this study is to show the success of the AutoLog System in removing lipids to less than 10mg/dl in vivo. The Autolog registry has two objectives:

1. to determine the lipid removal capabilities of the Medtronic AutoLog System.
2. to obtain in vivo data on blood component removal and washing capabilities of the Medtronic AutoLog System.

DETAILED DESCRIPTION:
Since the in house data strongly suggest that the Medtronic AutoLog is uniquely high performing in lipid removal in-vitro, the Registry AutoLog Lipid Removal and Blood Component Characterization is initiated to determine if the AutoLog system is successful in removing lipids in vivo as it is in-vitro. Therefore, it is expected that the lipid amounts after washing will be less than 10 mg/dl.

The study is designed as a multi-center, non-randomized, non-interventional, post market release study (a registry). The study has a single arm, without controls, as it is descriptive in nature.

ELIGIBILITY:
Inclusion Criteria:

* Patients with an indication for surgery procedures in which the hospital treatment protocol requires the routine use of an autotransfusion system are eligible for participation.

Exclusion Criteria:

* The use of citrate-based anticoagulant in patients with impaired liver function
* Gross contamination and/or septic procedures
* Surgery within the malignant area that may allow dissemination of tumor/malignant cells, if aspirated, into the autotransfusion system
* Caesarean sections in presence of amniotic fluid
* Presence of high concentrations of prostatic fluid
* Contamination of salvaged blood with drugs not intended for intravenous administration
* Use of collagen-based haemostatic agents and gel foam used in combination with any autotransfusion system
* Coagulopathy
* Not willing to sign a Patient Informed Consent/Data Release Form

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The subject population includes all subjects with an indication for cardiac surgery, orthopedic surgery etc. in which the hospital treatment protocol requires the routine use of an autotransfusion system, and who meet the inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 199 (Actual)
Dates: Start 2011-12; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
level of reduction of nonemulsified fat | after process
  The primary endpoint of this study is the level of reduction of nonemulsified fat after processing through the Medtronic AutoLog.

CONTACTS AND LOCATIONS:
Locations (6):
- Azienda Ospedaliera Universitaria Materdomini, Catanzaro, Italy
- Vilnius University Hospital Santariskiu Klinikos, Vilnius, Lithuania
- Institut national de chirurgie cardiaque et de cardiologie interventionnelle (INCCI), Luxembourg, Luxembourg
- VU Medisch Centrum, Amsterdam, Netherlands
- Zuid-Afrikaans Hospital, Pretoria, South Africa
- Universitetssjukhuset i Lund, Lund, Sweden